CLINICAL TRIAL: NCT00284960
Title: The Incidence and Treatment of Insulin Resistance Among Men With Erectile Dysfunction
Status: Completed | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 18805; NIH: K24 H001476
Record Dates: First submitted 2006-01-31; First posted 2006-02-01 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Erectile Dysfunction; Metabolic Syndrome; Insulin Resistance
Keywords: erectile dysfunction; metabolic syndrome; insulin resistance; etiology
MeSH Terms: conditions — Erectile Dysfunction; Metabolic Syndrome; Insulin Resistance

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Determine if men with erectile dysfunction (ED) are more likely to have insulin resistance compared to healthy controls.

DETAILED DESCRIPTION:
Insulin is a hormone produced by the body that lets sugar into the cells, where it is used for energy. Insulin resistance occurs when the body's cells have a decreased ability to react to insulin. This leads to an increase in insulin secretion. Over time, insulin resistance can lead to higher levels of sugar in the blood (diabetes), and can also contribute to obesity, high blood pressure, high cholesterol levels and heart disease. There are no simple tests to actually diagnose insulin resistance. Currently, the glucose tolerance test is used to diagnose IR, but it involves several blood draws over a 2-hour period. Another purpose of this study is to compare a blood test involving only one blood draw to the 2-hour glucose tolerance test, which involves several blood draws over a 2-hour period.

It is well known that diabetes often leads to erectile dysfunction. Because insulin resistance occurs before diabetes, it is possible that erectile dysfunction may occur in some individuals while they have insulin resistance, but before they develop diabetes. If this is true, it might be possible to use erectile dysfunction as a sign of insulin resistance, which may lead to more timely treatment of insulin resistance and may delay or prevent the development of diabetes, and the other problems mentioned above.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age, male,

Exclusion Criteria:

* diabetes, peyronies

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-06; Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J C Trussell, MD, Principal Investigator
Locations (1):
- Hershey Med Center, Hershey, Pennsylvania, United States